CLINICAL TRIAL: NCT06795672
Title: Tele-rehabilitation for Cognitive Disorders: a Randomized Controlled Trial in Patients with Stroke Outcomes
Brief Title: Tele-rehabilitation for Cognitive Disorders
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties in patient recruitment
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Valentina Varalta, Doctor, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3623CESC
Record Dates: First submitted 2025-01-21; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2022-03

CONDITIONS: Rehabilitation; Stroke; Telerehabilitation; Telemedicine
Keywords: stroke; telemedicine; rehabilitation
MeSH Terms: conditions — Stroke | interventions — Telerehabilitation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Telerehabilitation group (Experimental): Three hours of cognitive rehabilitation per week, performed remotely and independently, using a computerized device, which is pre-programmed based on the patient's needs.
  Interventions: Behavioral: Telerehabilitation
- In-person treatment (Active Comparator): Three hours of in-person cognitive rehabilitation per week using a computerized device.
  Interventions: Behavioral: Traditional in-person rehabilitation.

INTERVENTIONS:
Behavioral: Telerehabilitation — Three hours of cognitive rehabilitation per week, performed remotely and independently, using a computerized device, which is pre-programmed based on the patient's needs.
  Arms: Telerehabilitation group
Behavioral: Traditional in-person rehabilitation. — Three hours of in-person cognitive rehabilitation per week using a computerized device.
  Arms: In-person treatment

SUMMARY:
The aim of the study is to evaluate whether a computer-based cognitive treatment delivered via tele-rehabilitation produces an improvement in cognitive functioning comparable to the improvement achievable through the same treatment delivered in person in patients with stroke outcomes.

To investigate, using a custom-designed questionnaire, the feasibility and patient satisfaction with the rehabilitative treatment delivered via telemedicine compared to the same treatment delivered in person.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ischemic or hemorrhagic stroke;
* Age between 18 and 90 years;
* First stroke event;
* Stroke occurred more than 30 days ago;
* Adequate level of understanding;
* Presence of one or more of the following cognitive disorders:
* Memory disorders
* Attention disorders
* Executive function disorders
* Availability of an internet connection at the patient's home necessary for the telemedicine procedures.

Exclusion Criteria:

* Presence of other neurological disorders;
* Presence of pre-morbid cognitive decline;
* Psychiatric disorders in the medical history;
* Alcohol and/or drug abuse;
* Presence of severe uncorrected visual deficits.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Trail Making Test Part B (TMT-B) | From enrollment to the end of treatment and 2 months until the end of treatment
  Used as a measure of attentional set-shifting and mental flexibility. Time needed to complete the tasks is recorded.

SECONDARY OUTCOMES:
The Trail Making Test - A (TMT-A) | From enrollment to the end of treatment and 2 months until the end of treatment
  Used as a measure of psychomotor speed and visual search/attention skills
15 Words of Rey | From enrollment to the end of treatment and 2 months until the end of treatment
  To assess verbal learning ability and long-term verbal memory (IMMEDIATE RECALL: score ranging from 0 to 75. DELAYED RECALL: score ranging from 0 to 15).
Memory with interference - ENB 2 | From enrollment to the end of treatment and 2 months until the end of treatment
  to assess working memory through the memorization of letter triplets alongside a distracting task lasting 10 seconds in the first part and 30 seconds in the second. The maximum obtainable score is 9 for both parts of the test.
Dual task test | From enrollment to the end of treatment and 2 months until the end of treatment
  Dual Task to assess the ability to perform two tasks simultaneously (one verbal and one visuomotor)
Elithorn's Perceptual Maze Test | From enrollment to the end of treatment and 2 months until the end of treatment
  to investigate problem-solving abilities.
Stroop Test | From enrollment to the end of treatment and 2 months until the end of treatment
  to assess the speed and accuracy of automatic response inhibition.
Functional Independence Measure (FIM) | From enrollment to the end of treatment and 2 months until the end of treatment
  To evaluate the degree of disability.
Hospital Anxiety and Depression Scale | From enrollment to the end of treatment and 2 months until the end of treatment
  to assess the presence of depression and anxiety.
Short Form Health Survey 36 (SF-36) | From enrollment to the end of treatment and 2 months until the end of treatment
  to evaluate quality of life.
Feasibility, Satisfaction, and Cost Questionnaire | From enrollment to the end of treatment and 2 months until the end of treatment
  to assess the feasibility and satisfaction with the treatment and to evaluate the costs associated with it.

CONTACTS AND LOCATIONS:
Locations (1):
- Sezione medicina fisica e riabilitativa dipartimento di neuroscienze, Verona, verona, Italy